CLINICAL TRIAL: NCT01199315
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Modified-Release Formulations of AZD1446 in Young and Elderly Healthy Japanese Volunteers After Oral Single and Repeated Doses
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Modified-Release Formulations of AZD1446 After Oral Single and Repeated Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1950C00013
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: safety; tolerability; AZD1446; AD; ADHD; Japanese
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral capsule. Dose single and followed by 5-day repeated dosing. Specific doses depend on panel.
  Interventions: Drug: AZD1446
- 2 (Placebo Comparator): Oral capsule. Dose single and followed by 5-day repeated dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — oral capsule, Moderate Release
  Arms: 1
Drug: Placebo — oral capsule
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety, tolerability and pharmacokinetics of AZD1446 in young and elderly healthy Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese volunteers, aged ≥20 to ≤50 years for male young volunteers, ≥65 to ≤80 years for male or post-menopausal female elderly volunteers.
* BMI between 18 and 27 kg/m2 and weigh at least 50 kg and no more than 90 kg (for the elderly female, weigh at least 45 kg and no more than 90 kg).

Exclusion Criteria:

* History of severe allergy/hypersensitivity reactions including drug-allergy or drug hypersensitivity reactions, or ongoing allergy/hypersensitivity.
* History or present symptoms or signs of Quincke oedema, angiooedema, or urticaria pigmentosa, or history of repeated episodes of urticaria.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of AZD1446 following single and repeated doses of an orally administered MR capsule of AZD1446 in healthy young and elderly Japanese volunteers by adverse events, vital signs, laboratory variables and ECG. | During the whole study period, ca. 50 days

SECONDARY OUTCOMES:
To determine PK of AZD1446 following single and repeated doses of AZD1446 MR capsule in healthy young and elderly Japanese volunteers. | PK samplings are taken at defined timepoints during residential period, 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, Study Director — AstraZeneca R&D Södertälje; Shunji Matsuki, PhD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Fukuoka, Japan